CLINICAL TRIAL: NCT02251600
Title: A Multi-center Study to Evaluate the Pharmacokinetics of 21-Desacetyldeflazacort and the Safety of Deflazacort After Oral Administration of Deflazacort Tablets to Children and Adolescent Subjects With Duchenne Muscular Dystrophy
Brief Title: A Pharmacokinetic Study of Oral Deflazacort in Children and Adolescent Subjects With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MP-104-CL-005
Record Dates: First submitted 2014-09-22; First posted 2014-09-29 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Pediatric; Adolescent; Deflazacort
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deflazacort (Experimental): This is an open label and single period study , dosed with 0.9mg/kg Deflazacort.
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort — Oral deflazacort administered once daily at 0.9 mg/kg for eight days
  Other Names: DFZ

SUMMARY:
Study to characterize the single-state and steady-state dosing of oral deflazacort in pediatric and adolescents subjects.

DETAILED DESCRIPTION:
This is an open label, single period study in 24 male DMD subjects consisting of children (ages 4-12, inclusive) and adolescents (ages 13-16, inclusive) with at least 12 subjects between the ages of 4-12 (children). Subjects taking maintenance corticosteroid therapy will be required to take their dose of corticosteroid 24 hours (± 2 hours) prior to the first dose of deflazacort on Day 1. Subjects receiving deflazacort as maintenance corticosteroid therapy must take their last dose at least 30 days prior to the first dose of deflazacort on Day 1. Concomitant corticosteroid therapy will be prohibited during the study while the subject is taking deflazacort. On Day 1, a single oral dose of deflazacort under fasting conditions will be administered in the CRU followed by blood sampling for plasma analysis of DFZ and 21-desacetyl-DFZ for 8 hours. Following the 8 hour PK sample on Day 1, subjects will be given medication to take at home for once-daily, morning dosing on Days 2 through 7 (+2 days). On Day 8 (+2 days), subjects will return for a PK sample predose and an 8th oral dose of deflazacort under fasting conditions which will be administered in the CRU followed by PK sampling for 8 hours.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations on Days 1 and 8 (+2 days). Subjects will be contacted via telephone approximately 7 days (± 1 day) following study drug administration on Day 8 (+2 days) for a follow-up assessment to determine if any adverse event (AE) has occurred since the last study visit. Subjects who terminate the study early will be contacted if the Principal Investigator (PI) deems necessary.

Subjects that complete this study or receive at least one dose of study medication will be eligible for an open-label extension study with deflazacort treatment conducted under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
* The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* If above the age of 7, the subject signs and dates a written, informed assent form (IAF) and any required privacy authorization prior to the initiation of any study procedures.
* The subject must have confirmed diagnosis of Duchenne Muscular Dystrophy defined as muscle biopsy and dystrophin analyses consistent with DMD or DNA mutation and analysis by PCR or Southern blot techniques to detect gene deletions as well as:

  1. onset of weakness before 5 years of age;
  2. proximal muscle weakness;
  3. increased serum creatine kinase more than 10 times the upper limit of normal (ULN);
* The subject is male and aged 4 to 16 years, inclusive.
* The subject weighs at least 13 kg and has a Body Mass Index (BMI) of ≤ 40.
* Willingness and ability to comply with scheduled visits, oral drug administration, and study procedures including blood sample draws (total blood volume collected not to exceed 50 mL for the study duration or 25 mL on any single study day [≤ 3 mL/kg])
* The subject has a life expectancy of >1 year.
* Up to date on all childhood vaccinations, specifically varicella vaccine (chicken pox).
* Baseline health is judged to be stable based on medical history, physical examination, laboratory profiles, vital signs, or ECGs at screening, as deemed by the Investigator.
* Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose.
* The subject is able to take tablets.

Exclusion Criteria:

* The subject has received any investigational compound and/or has participated in another clinical study within 90 days prior to study treatment with the exception of observational cohort studies or non-interventional studies.
* The subject has received deflazacort within 30 days or previous discontinued deflazacort due to an intolerable reaction.
* The subject is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g. spouse, parent, child, sibling) or may consent under duress.
* Any significant finding on the Columbia suicide severity rating scale (C SSRS) for subjects (ages 12-16, inclusive), in the opinion of the PI, warrants exclusion from this study.
* The subject has, in the judgment of the investigator, clinically significant abnormal clinical chemistry laboratory parameters that may affect safety at Screening.
* The subject has, in the judgment of the investigator, a history or current medical condition that could affect safety including, but not limited to:

  1. Major renal or hepatic impairment
  2. Immunosuppression or other contraindications for corticosteroid treatment
  3. History of chronic systemic fungal or viral infections
  4. Diabetes mellitus
  5. Idiopathic hypocalcuria
  6. Symptomatic cardiomyopathy at screening
* The subject has a history of hypersensitivity or allergic reaction to steroids or their formulations including, but not limited to lactose, sucrose, etc.
* Inability to take tablets as assessed by site investigator.
* Unable to refrain from or anticipates the use of:

  * Any medications at least 4 hours before and after dosing on PK Days 1 and 8.
  * Any vitamins, vitamins with minerals, and/or meal supplementation (e.g., Ensure, Boost, etc.) at least 4 hours before and after dosing on PK Days 1 and 8.
  * Any drug, including prescription and non prescription medications, and herbal remedies known to be significant inhibitors of CYP 3A4 enzymes and/or P gp for 14 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of pharmacokinetic/pharmacodynamic interaction with study drug. Acetaminophen may be permitted during the study (doses to be based upon appropriate age/weight ranges.
  * Any drugs known to be significant inducers of CYP 3A4 enzymes and/or P gp for 28 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics interaction with study drug.
* Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* Positive urine drug or alcohol results at screening or check in.
* Positive urine cotinine at screening.
* Positive results at screening for HIV, HBsAg, or HCV.
* Hemoglobin level below the lower limit of normal at screening.
* Donation of blood or significant blood loss within 56 days prior to the first dose of study drug.

Ages: 4 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration time curve, from time 0 to the last measurable concentration non-zero, for single-state pharmacokinetics on Day 1 of deflazacort and 21-desacetyl-DFZ, the active metabolite | Day 1, Day 8
  The area under the plasma concentration time curve, from time 0 to the last measurable concentration non-zero, for single-state pharmacokinetics on Day 1 of deflazacort and 21-desacetyl-DFZ, the active metabolite
The area under the plasma concentration versus time curve over the final dosing interval for steady state pharmacokinetics on Day 8 of deflazacort and 21-desacetyl-DFZ, the active metabolite | Day 8
  The area under the plasma concentration versus time curve over the final dosing interval for steady state pharmacokinetics on Day 8 of deflazacort and 21-desacetyl-DFZ, the active

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Day 1-8
  To assess the safety and tolerability of single-dose and steady-state deflazacort in DMD subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Smith, MD, Study Chair — Drug Safety Solutions/Celerion
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Rochester Medical Center, Rochester, New York
  - University of Utah, Salt Lake City, Utah